CLINICAL TRIAL: NCT00628186
Title: Prospective, Randomized, and Controlled Trial That Lost Stent Versus External Stent of Pancreaticojejunostomy After Pancreaticoduodenectomy
Brief Title: Randomized Controlled Trial on Pancreatic Stent Tube in Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP-0501
Record Dates: First submitted 2008-01-23; First posted 2008-03-04 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer; Ampullary Cancer; Pancreatitis; Duodenal Cancer
Keywords: pancreaticoduodenectomy; stent; pancreaticojejunostomy; hospital stay; complication; pancreatic fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms; Pancreatitis; Duodenal Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Pancreaticojejunostomy has a risk factor of pancreatic fistula. Type of stent tube (external stent vs. short stent)across pancreaticojejunostomy was randomized for the patients with pancreaticoduodenectomy.
  Interventions: Device: external drainage tube [polyethylene pancreatic drainage tube]; Device: internal drainage tube [polyethylene pancreatic drainage tube]

INTERVENTIONS:
Device: external drainage tube [polyethylene pancreatic drainage tube] — External drainage tube was intubated with a 5F polyethylene pancreatic drainage tube with a small knob (Sumitomo Bakelite Co., Japan)(MD41515) across pancreaticojejunostomy in pancreaticoduodenectomy, and exteriorized through the jejunal limb.
  Other Names: polyethylene pancreatic drainage tube(S/N MD41515)
Device: internal drainage tube [polyethylene pancreatic drainage tube] — Internal drainage tube was intubated 5cm length of stent tube cut a 5F polyethylene pancreatic drainage tube with a small knob across pancreaticojejunostomy in pancreaticoduodenectomy, and pancreatic juice was led to reconstructed jejunum.
  Other Names: polyethylene pancreatic drainage tube(S/N MD41515)

SUMMARY:
The purpose of this study is to determine which stent type is effective in the decrease of postoperative stay and complications across pancreaticojejunostomy after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
This study compared the postoperative hospital stay and complications of lost stent with external stent after pancreaticoduodenectomy. The complications of pancreaticoduodenectomy are important to affect the postoperative course, and, a stent tube often places across pancreaticojejunostomy to reduce complications. However, there is no report that demonstrates the postoperative course between pancreatic stent types. We conducted a prospective randomized trial on 100 patients who underwent pancreaticoduodenectomy comparing external stent and lost stent.

The primary endpoint was defined as postoperative hospital stay. The secondary endpoints were mortality and morbidity, including pancreatic fistula, delayed gastric emptying, intra-abdominal hemorrhage, and intra-abdominal abscess. Patients were recruited into this study before surgery, on the basis of whether pancreatic head resection was anticipated at WMUH for pancreatic head and periampullary disease, and appropriate informed consent was obtained. Exclusion criteria was 1) patients with severe complications which were possible to prolong hospital stay, 2) patients who were diagnosed inadequacy for this study by a physician, 3) patients who could not be placed a pancreatic stent tube, and 4) patients without an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* On the basis of whether pancreatic head resection was anticipated at WMUH for pancreatic head and periampullary disease, and appropriate informed consent was obtained.

Exclusion Criteria:

* Patients with severe complications which were possible to prolong hospital stay
* Patients who were diagnosed inadequacy for this study by a physician
* Patients who could not be placed a pancreatic stent tube
* Patients without an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-04; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
the length of hospital stay after pancreaticoduodenectomy | the day of discharge

SECONDARY OUTCOMES:
early and late complications after pancreaticoduodenectomy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Masaji Tani, MD, Study Director — Wakayama Medical University, Second Department of Surgery
Locations (1):
- Wakayama Medical University , Second Department of Surgery, 811-1 Kimiidera, Wakayama, Wakayama, Japan

REFERENCES:
- [Background] Tani M, Kawai M, Terasawa H, Ina S, Hirono S, Shimamoto T, Miyazawa M, Uchiyama K, Yamaue H. Prognostic factors for long-term survival in patients with locally invasive pancreatic cancer. J Hepatobiliary Pancreat Surg. 2007;14(6):545-50. doi: 10.1007/s00534-007-1209-6. Epub 2007 Nov 30. PMID 18040618
- [Background] Kawai M, Tani M, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Shimamoto T, Yamaue H. CLIP method (preoperative CT image-assessed ligation of inferior pancreaticoduodenal artery) reduces intraoperative bleeding during pancreaticoduodenectomy. World J Surg. 2008 Jan;32(1):82-7. doi: 10.1007/s00268-007-9305-y. PMID 18027017
- [Background] Kawai M, Tani M, Terasawa H, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Yamaue H. Early removal of prophylactic drains reduces the risk of intra-abdominal infections in patients with pancreatic head resection: prospective study for 104 consecutive patients. Ann Surg. 2006 Jul;244(1):1-7. doi: 10.1097/01.sla.0000218077.14035.a6. PMID 16794381
- [Background] Terasawa H, Uchiyama K, Tani M, Kawai M, Tsuji T, Tabuse K, Kobayashi Y, Taniguchi K, Yamaue H. Impact of lymph node metastasis on survival in patients with pathological T1 carcinoma of the ampulla of Vater. J Gastrointest Surg. 2006 Jun;10(6):823-8. doi: 10.1016/j.gassur.2006.01.013. PMID 16769538
- [Background] Tani M, Kawai M, Terasawa H, Ina S, Hirono S, Uchiyama K, Yamaue H. Does postoperative chemotherapy have a survival benefit for patients with pancreatic cancer? J Surg Oncol. 2006 May 1;93(6):485-90. doi: 10.1002/jso.20440. PMID 16615151
- [Background] Tani M, Terasawa H, Kawai M, Ina S, Hirono S, Uchiyama K, Yamaue H. Improvement of delayed gastric emptying in pylorus-preserving pancreaticoduodenectomy: results of a prospective, randomized, controlled trial. Ann Surg. 2006 Mar;243(3):316-20. doi: 10.1097/01.sla.0000201479.84934.ca. PMID 16495694
- [Background] Tani M, Kawai M, Terasawa H, Ueno M, Hama T, Hirono S, Ina S, Uchiyama K, Yamaue H. Complications with reconstruction procedures in pylorus-preserving pancreaticoduodenectomy. World J Surg. 2005 Jul;29(7):881-4. doi: 10.1007/s00268-005-7697-0. PMID 15951940
- [Background] Tani M, Onishi H, Kinoshita H, Kawai M, Ueno M, Hama T, Uchiyama K, Yamaue H. The evaluation of duct-to-mucosal pancreaticojejunostomy in pancreaticoduodenectomy. World J Surg. 2005 Jan;29(1):76-9. doi: 10.1007/s00268-004-7507-0. PMID 15592915
- [Background] Kawai M, Uchiyama K, Tani M, Onishi H, Kinoshita H, Ueno M, Hama T, Yamaue H. Clinicopathological features of malignant intraductal papillary mucinous tumors of the pancreas: the differential diagnosis from benign entities. Arch Surg. 2004 Feb;139(2):188-92. doi: 10.1001/archsurg.139.2.188. PMID 14769579
- [Background] Yamaue H, Tani M, Onishi H, Kinoshita H, Nakamori M, Yokoyama S, Iwahashi M, Uchiyama K. Locoregional chemotherapy for patients with pancreatic cancer intra-arterial adjuvant chemotherapy after pancreatectomy with portal vein resection. Pancreas. 2002 Nov;25(4):366-72. doi: 10.1097/00006676-200211000-00008. PMID 12409831
- [Derived] Tani M, Kawai M, Hirono S, Ina S, Miyazawa M, Shimizu A, Yamaue H. A prospective randomized controlled trial of internal versus external drainage with pancreaticojejunostomy for pancreaticoduodenectomy. Am J Surg. 2010 Jun;199(6):759-64. doi: 10.1016/j.amjsurg.2009.04.017. Epub 2010 Jan 15. PMID 20074698